CLINICAL TRIAL: NCT00650390
Title: Open Label Study to Assess Efficacy and Safety of the Fully Human Anti-TNF-Alpha Monoclonal Antibody Adalimumab
Acronym: PROWD
Status: Approved for marketing | Type: Expanded Access
Sponsor: Abbott (Industry)
Responsible Party: Lawrence McNamee, Abbott
Other Study IDs: M02-532
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2008-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

INTERVENTIONS:
Biological: adalimumab — 40 mg adalimumab every other week
  Other Names: ABT-D2E7; Humira

SUMMARY:
The study was to explore the efficacy of adalimumab in subjects previously treated with infliximab and failed infliximab treatment due to lack of efficacy or intolerance. To explore the safety of adalimumab in subjects previously treated with infliximab.

ELIGIBILITY:
Inclusion Criteria:

* Males and females >= 18 years of age
* ACR criteria for RA diagnosis for at least 6 months
* Active RA defined as a DAS 28 >3.2 at study entry
* Unsatisfactory response, loss of response or intolerance to prior infliximab treatment
* A negative pregnancy test for females of childbearing potential

Exclusion Criteria:

* Patient who had previous treatment with cyclophosphamide and chlorambucil
* Treatment within the last 8 weeks with infliximab
* Prior treatment with more than one DMARD or DMARD combination following infliximab treatment
* Prior treatment with biologics (Investigational or Commercial) RA therapies other than infliximab
* History of cancer, other than successfully treated squamous cell or basal cell carcinoma or lymphoproliferative disease
* Prior treatment with total lymphoid irradiation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

REFERENCES:
- [Derived] Burmester GR, Landewe R, Genovese MC, Friedman AW, Pfeifer ND, Varothai NA, Lacerda AP. Adalimumab long-term safety: infections, vaccination response and pregnancy outcomes in patients with rheumatoid arthritis. Ann Rheum Dis. 2017 Feb;76(2):414-417. doi: 10.1136/annrheumdis-2016-209322. Epub 2016 Jun 23. PMID 27338778